CLINICAL TRIAL: NCT01942551
Title: Safety and Pharmacokinetic Interaction Study of Tadalafil and Dutasteride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dongkook Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: DK-DT-001
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Benign Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tadalafil; Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tadalafil, dutasteride (Experimental)
  Interventions: Drug: Tadalafil; Drug: Dutasteride
- dutasteride, tadalafil (Experimental)
  Interventions: Drug: Tadalafil; Drug: Dutasteride

INTERVENTIONS:
Drug: Tadalafil
Drug: Dutasteride

SUMMARY:
This is an open-label, two-arm, one-sequence, cross-over study to evaluate the safety and pharmacokinetic interaction after oral concomitant administration of tadalafil and dutasteride in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 20 to 29 years 2. Weight 60 kg or more, within 20% of Ideal body weight 3. No congenital or chronic diseases, no disease symptoms or findings 4. Eligible according to the laboratory results of hematology, blood chemistry and urinalysis 5. Voluntarily signed the informed consent form

Exclusion Criteria:

* 1. Clinically significant disorders of hepatobiliary system, kidney, neurology, respiratory, hemato-oncology, endocrine, dermatology, urology, ophthalmology, psychiatry, musculo-skeletal system, immunology, otorhinolaryngology, and cardiovascular system 2. Gastrointestinal diseases or surgery which may affect absorption of the investigational products 3. hypersensitivity to tadalafil or phosphodiesterase type 5 inhibitor, and dutasteride or 5-α reductase inhibitor 4. Lactose intolerance 5. SBP ≥ 140 mmHg or < 90 mmHg or DBP ≥ 95 mmHg or < 60 mmHg 6. Serum creatinine > ULN 7. History or positive result of drug abuse 8. Drugs which induce or inhibit drug metabolism including barbiturates within 1 month 9. Prescribed drugs or herbal medicines within 2 weeks, or over-the counter drugs or vitamins within 1 week 10. CYP3A4 inhibitors or CYP3A4 inducers within 2 weeks 11. Food including grapefruit from Week -1 to final dose 12. Participated and administered the investigational products in other clinical trial within 2 months 13. Donated whole blood within 2 months or apheresis within 1 month, or transfusion within 1 month 14. Plans to donate blood for at least 6 months after final dose of dutasteride 15. Scheduled dental treatment and elective surgery from informed consent to post-study visit 16. Excessive alcohol consumption (> 21 units/week, 1 unit = 10 g of pure alcohol) 17. Smoked more than 10 cigarettes a day for past 3 months 18. Not eligible due to other reasons including laboratory results

Ages: 20 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) of tadalafil | 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24 h
Cmax of tadalafil | 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24 h
Area Under Curve (AUC) of dutasteride | 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, 48, 72, 96, 144, 192, 240, 288, 336 h
Cmax of dutasteride | 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, 48, 72, 96, 144, 192, 240, 288, 336 h

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea